CLINICAL TRIAL: NCT00722384
Title: An Open Label Study for the Evaluation of Tolerability of Five Dose Levels of Cand5 by Single Intravitreal Injection in Patients With Wet Age-Related Macular Degeneration
Brief Title: Open Label Study for the Evaluation of Tolerability of Five Dose Levels of Cand5
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Denis O'Shaughnessy, Opko Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACU101
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2008-07-25 (Estimated); Status verified 2008-07

CONDITIONS: Macular Degeneration
Keywords: AMD; Macular Degeneration; Opko Health; Acuity Pharmaceuticals; bevasiranib; Cand5; Age-Related
MeSH Terms: conditions — Macular Degeneration | interventions — bevasiranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): 0.1 mg bevasiranib in the study eye
  Interventions: Drug: bevasiranib
- 2 (Experimental): 0.33 mg bevasiranib in the study eye,
  Interventions: Drug: bevasiranib
- 3 (Experimental): 1.0 mg bevasiranib in the study eye
  Interventions: Drug: bevasiranib
- 4 (Experimental): 1.5 mg bevasiranib in the study eye
  Interventions: Drug: bevasiranib
- 5 (Experimental): 3.0 mg bevasiranib in the study eye.
  Interventions: Drug: bevasiranib

INTERVENTIONS:
Drug: bevasiranib
  Other Names: Cand5
Drug: bevasiranib — The first three patients enrolled will receive 0.1 mg Cand5 in the study eye, the next three patients enrolled will receive 0.33 mg Cand5 in the study eye, the following three patients enrolled will receive 1.0 mg Cand5 in the study eye, the following three patients enrolled will receive 1.5 mg Cand5 in the study eye, and the remaining three patients enrolled will receive 3.0 mg Cand5 in the study eye. The third patient enrolled at each dose level will complete their two-week visit before the next dose level group may be treated.

SUMMARY:
To establish the tolerability and preliminary efficacy of Cand5 by a single intravitreal injection in patients with wet age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Patients with subfoveal predominantly classic, minimally classic and purely occult lesions, secondary to age related macular degeneration, with a total lesion size (including blood, atrophy/scar and neovascularization) of < 12 total disc areas, of which at least 50% are active CNV.
* Patients must have visual acuity 20/50 to 20/320 in the study eye.
* Patients must have better visual acuity in the fellow eye than the study eye.
* Subretinal hemorrhage (if any) must comprise no more than 50% of total lesion size.

Exclusion Criteria:

* Patients with concomitant eye disease, including glaucoma, uveitis, diabetic retinopathy, presence of pigment epithelial tears or rips, acute ocular or periocular infection in the study eye.
* Patients with > 3 prior PDT treatments with Visudyne in the study eye.
* Patients who received PDT in the study eye within eight weeks prior to the baseline angiography/photography.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-08; Primary Completion 2007-08 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Complications, including those related to the intravitreal injection, and adverse events, and loss of lines of best-corrected visual acuity, slit lamp findings, lens opacification, intraocular pressure, fundus findings, and laboratory findings.

SECONDARY OUTCOMES:
Stabilization of visual acuity (prevention of loss of three or more lines on the ETDRS chart), stabilization of lesion size, lack of leakage of lesion, or decrease in subretinal fluid

CONTACTS AND LOCATIONS:
Locations (1):
- OPKO site, Morristown, New Jersey, United States